CLINICAL TRIAL: NCT03683797
Title: Testing the Efficacy of a Post-discharge Call Program on the Rate of Readmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RCT post-discharge calls
Record Dates: First submitted 2018-08-28; First posted 2018-09-25 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Care Transitions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-discharge call (Experimental): Patients in this arm will receive a call from a clinical care coordinator after they have been discharged from NYU Langone Health.
  Interventions: Other: Post-discharge call
- No post-discharge call (No Intervention): Patients in this arm will not receive a call from a clinical care coordinator after they have been discharged from NYU Langone Health.

INTERVENTIONS:
Other: Post-discharge call — Patients will receive a call 1-3 days after they were discharged from the hospital to make sure their healthcare needs are being met.
  Arms: Post-discharge call

SUMMARY:
NYU Langone Health patients receive a call from a clinical care coordinator after they are discharged from the hospital (within 1-3 days). The current study is testing the efficacy of this program.

ELIGIBILITY:
Inclusion Criteria:

* All patients discharged from NYU Langone Health who are eligible to receive a call from a clinical care coordinator after they were discharged from the hospital.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3267 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Rate of readmission | 6 months
  Number of patients admitted to a hospital within after being discharged from an earlier hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, MHS, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States